CLINICAL TRIAL: NCT05907863
Title: Intracardiac Echocardiography Guided vs. Electroanatomical Mapping System Guided Slow Pathway Ablation in Patients With Atrioventricular Nodal Reentrant Tachycardia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Peter Kupo MD, PhD, assistant professor, University of Pecs
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UPEP2023/1
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Heart Rhythm Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracardiac echo guided ablation (Experimental)
  Interventions: Other: Use of intracardiac echocardiography
- Standard, electroanatomical mapping system guided ablation (No Intervention)

INTERVENTIONS:
Other: Use of intracardiac echocardiography — intracardiac echocardiography guided slow pathway ablation in patients with AVNRT
  Arms: Intracardiac echo guided ablation

SUMMARY:
Study protocol

To prepare for the electrophysiologic study, antiarrhythmic drugs were discontinued at least five half-lives before the procedure and were under conscious sedation using midazolam ± fentanyl while fasting.

ICE-guided ablation group In patients randomized to ICE-guided ablation group, catheter placement was initially performed using fluoroscopy guidance, after local anesthesia. A decapolar steerable catheter was placed in the coronary sinus (CS), a quadripolar electrode catheter was positioned in the right ventricular apex and an ablation catheter was inserted to record the His bundle electrogram. Twelve-lead electrocardiogram and intracardiac electrograms were recorded and saved on a digital recording system using a band pass filter of 30 to 500 Hz. Electrical stimulation techniques were used to test atrioventricular nodal conduction and induce AVNRT, with the S2 coupling interval being gradually shortened after each drive-train until tachycardia was induced, AV conduction block occurred, or the atrial refractory period was reached. If tachycardia was not inducible, isoprenaline infusion was given to increase the heart rate by at least 20%, and the same stimulation protocol was repeated during both the infusion and washout phases. The diagnosis of AVNRT was made using established electrophysiologic criteria and pacing maneuvers. This involved assessing the A-(H)-V response after ventricular overdrive pacing, with an SA-VA interval greater than 85 ms, and a corrected postpacing interval minus tachycardia cycle length greater than 110 ms.

After confirmation of the diagnosis of AVNRT through the diagnostic EP study, the quadripolar electrode catheter was removed and replaced with an 8F ICE catheter for mapping and SP ablation. The echo-transducer was positioned in the low right atrium at the 6 o'clock position and rotated clockwise towards the septum to allow for visualization of the anatomic landmarks. The proximity of the ablation catheter to the compact AV node was determined by the distance from the aortic valve, which marks the recording site of a proximal His potential. In cases of ineffective ablation, the catheter was moved closer to the aortic valve, but always maintaining a distance of at least 0.5 cm, and RF application was attempted again. RF energy was delivered starting just below the CS with a power output of 30 W and a preset temperature of 55°C. Effective applications were continued for 30 to 60 s and considered successful when junctional rhythm appeared. RF application was immediately halted if there was catheter displacement, sudden impedance rise, prolongation of PR interval, anterograde AV or retrograde VA block.

Electroanatomical mapping system -guided ablation group An ablation catheter was inserted into the heart to create an anatomical map by CARTO of the right atrium after local anesthesia, and the location of the His bundle was tagged. Decapolar and quadripolar diagnostic catheters were positioned thereafter into appropriate position as described above. After confirming the diagnosis of AVNRT, mapping of the slow pathway was started by NAVISTAR catheter guided by EAMS and aiming at an atrial-to-ventricular electrogram amplitude ratio of 1:3-1:5. If the ablation endpoint was not reached after 8 radiofrequency (RF) applications, patients in the EMAS-guided ablation group were allowed to crossover to an ICE-guided procedure.

The ablation procedure was deemed successful if, following a 20-minute waiting period, the arrhythmia failed to be induced and there were no instances of more than one echo beat observed, both in the presence and absence of isoprenaline.

The procedure time was measured from the initial femoral puncture until the withdrawal of the catheters. The mapping plus ablation time was calculated from the start of the SP mapping until the end of the last attempted ablation. Fluoroscopy time, radiation dose, and dose-area product (DAP) were automatically recorded by the fluoroscopy system. The ablation data, including the total number of RF applications, sum of delivered RF energy in Watts, and the total ablation time in seconds, were calculated and stored by the EP recording system (CardioLab, GE Healthcare).

ELIGIBILITY:
Inclusion Criteria:

patients with documented paroxysmal supraventricular tachycardias

Exclusion Criteria:

* redo procedures
* pregnancy
* age under 18
* other arrhythmias in addition to AVNRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
procedural time | during the procedure

SECONDARY OUTCOMES:
ablation time | during the procedure
fluoroscopy useage | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pecs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No